CLINICAL TRIAL: NCT01083758
Title: Effect of Calcipotriol Plus Betamethasone Dipropionate Topical Suspension on the HPA Axis and Calcium Metabolism in Adolescent Subjects (Aged 12 to 17 Years) With Scalp Psoriasis
Brief Title: Safety and Efficacy of LEO 80185 Topical Suspension in Adolescent Subjects (Aged 12 to 17) With Scalp Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBL 0801; 2008-007606-11 (EudraCT Number)
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2015-08

CONDITIONS: Scalp Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEO 80185 (Taclonex® Scalp topical suspension/ Xamiol® gel) (Other)
  Interventions: Drug: LEO 80185 (Taclonex® Scalp topical suspension/Xamiol® gel)

INTERVENTIONS:
Drug: LEO 80185 (Taclonex® Scalp topical suspension/Xamiol® gel) — Topical suspension applied once daily for up to 8 weeks
  Other Names: LEO 80185 topical suspension

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of once daily use of LEO 80185 topical suspension in adolescent subjects (aged 12 to 17 years) with scalp psoriasis. LEO 80185 topical suspension has marketing approval in many countries under the brand names Taclonex Scalp® Topical Suspension and Xamiol® gel for the treatment of scalp psoriasis in adults. No studies have been performed in subjects younger than 18 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent given by parent(s) or legal guardian following their receipt of verbal and written information about the study
* Subjects will receive verbal and written information and will provide written assent to the study
* Any race or ethnicity
* Clinical signs of psoriasis vulgaris on trunk and/or limbs, or earlier diagnosed with psoriasis vulgaris on trunk and/or limbs
* At Screening Visit 2 and Visit 1 a clinical diagnosis of scalp psoriasis which is:

  * amenable to topical treatment with a maximum of 60 g of study medication per week, and
  * of an extent of more than or equal to 20% of the scalp area
  * of at least moderate severity according to the investigator's global assessment
* Subjects with a normal HPA axis function at SV2 including serum cortisol concentration above 5 mcg/dl before ACTH challenge and serum cortisol concentration above 18 mcg/dl 30 minutes after ACTH challenge
* A serum albumin-corrected calcium below the upper reference limit at Screening Visit 2
* Females of child-bearing potential must have a negative urine pregnancy test result and must agree to use a highly effective method of contraception (abstinence is an acceptable method).

Exclusion Criteria (summary):

* A history of serious allergy, allergic asthma or serious allergic skin rash
* Known or suspected hypersensitivity to any medication (including ACTH/cosyntropin/tetracosactide) or to any component of the LEO 80185 topical suspension or CORTROSYN
* Systemic treatment with corticosteroids (including inhaled and nasal steroids) within 12 weeks prior to Screening Visit 2 or during the study
* Topical treatment with corticosteroids within 2 weeks prior to Screening Visit 2 or during the study
* Oestrogen therapy (including contraceptives) or any other medication known to affect cortisol levels or HPA axis integrity within 4 weeks prior to Screening Visit 2 or during the study
* Enzymatic inductors (e.g., barbiturates, phenytoin, rifampicin)or cytochrome P450 inhibitors (e.g., ketoconazole, itraconazole, metronidazole) within 4 weeks prior to Screening Visit 2 or during the study. Topical ketoconazole 2 weeks prior to Screening Visit 2
* Hypoglycemic sulfonamides or Antidepressive medications within 4 weeks prior to Screening Visit 2 or during the study
* Known or suspected endocrine disorder that may affect the results of the ACTH challenge test
* Systemic treatment with biological therapies (marketed or not marketed), with a possible effect on scalp psoriasis within the following time period prior to Visit 1 and during the study within 4 weeks/5 half-lives (whichever is longer) prior to Visit 1
* Systemic treatment with therapies other than biologicals, with a possible effect on scalp psoriasis (e.g., retinoids, immunosuppressants, PUVA) within 4 weeks prior to Visit 1 (Day 0) or during the study
* Planned initiation of, or changes to, concomitant medication that could affect scalp psoriasis (e.g., betablockers, chloroquine, lithium, ACE inhibitors) during the study
* Other inflammatory skin diseases that may confound the evaluation of scalp psoriasis
* Known or suspected disorders of calcium metabolism associated with hypercalcaemia

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence F Eichenfield, MD, Principal Investigator — Rady Children's Hospital, San Diego
Locations (6):
- United States (6):
  - Rady Children's Hospital San Diego, San Diego, California
  - Leavitt Medical Associates of Florida, Inc., Jacksonville, Florida
  - Leavitt Medical Associates of Florida, Inc., Ormond Beach, Florida
  - Peachtree Dermatology Associates, PC, Atlanta, Georgia
  - Deaconess Clinic, Evansville, Indiana
  - Skin Specialists, PC, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start date: 12 April 2010 Completion date: 8 August 2012
Pre-assignment Details: Prior to Visit 1 (Day 0), a wash-out period (up to 8 weeks, as defined by the exclusion criteria) was to be completed if the subject had been treated with antipsoriatic treatments or other relevant medication; 2 screening visits were planned.
Groups:
- LEO 80185 Gel: Taclonex® Scalp Topical Suspension/Daivobet® gel /Dovobet® gel/Xamiol® gel Calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate) gel once daily for up to 8 week to treat psoriasis on the scalp
Period: Overall Study
Arm/Group | LEO 80185 Gel
Started | 31
Completed | 29
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Adverse Drug Reactions (ADRs)
Description: Adverse events for which the investigator did not describe the causal relationship to IP as not related
Time Frame: Throughout trial, up to 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 31
percentage of participants | 3.2

2. Primary Outcome: Subjects With Serum Cortisol Concentration of ≤18 mcg/dl at 30 Minutes After ACTH-challenge at Week 4
Description: Adrenal function can be measured by injecting a synthetic subunit of ACTH (Adrenocorticotropic hormone), and then measure the production of cortisol by the adrenal glands in response to this at 30 minutes after the injection.
Time Frame: Week 4
Population: Per Protocol Population (based on the Full Analysis Set, but excluding subjects who did not apply any study medication, meet the inclusion criterion concerning adrenal function at baseline, or provide any results for the ACTH-challenge test after receiving study treatment)
Measure: Number; unit: participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 30
participants | 1

3. Secondary Outcome: Change in Plasma PTH From Baseline (SV2) to Week 4 and Week 8
Description: Change in plasma PTH (parathyroid hormone) from Baseline (SV2 = screening visit 2) to Week 4 and Week 8
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 27
ng/L | -3.2 (15.6)

4. Primary Outcome: Subjects With Serum Cortisol Concentration of ≤18 mcg/dl at 30 Minutes After ACTH-challenge at Week 8
Description: Adrenal function can be measured by injecting a synthetic subunit of ACTH Adrenocorticotropic hormone), and then measure the production of cortisol by the adrenal glands in response to this at 30 minutes after the injection.
Time Frame: week 8
Population: Per Protocol Population
Measure: Number; unit: participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 26
participants | 0

5. Primary Outcome: Subjects With Serum Cortisol Concentration of ≤18 mcg/dl at 30 and 60 Minutes After ACTHchallenge at Week 4.
Description: Adrenal function can be measured by injecting a synthetic subunit of ACTH Adrenocorticotropic hormone), and then measure the production of cortisol by the adrenal glands in response to this at 30 and 60 minutes after the injection.
Time Frame: week 4
Population: Per Protocol Population
Measure: Number; unit: participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 29
participants | 0

6. Primary Outcome: Subjects With Serum Cortisol Concentration of ≤18 mcg/dl at 30 and 60 Minutes After ACTH-challenge at Week 8.
Description: Adrenal function can be measured by injecting a synthetic subunit of ACTH (Adrenocorticotropic hormone), and then measure the production of cortisol by the adrenal glands in response to this at 30 and 60 minutes after the injection.
Time Frame: week 8
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 25
participants | 0

7. Primary Outcome: Change in Albumincorrected Serum Calcium From Baseline (SV2) to Week 4, Week 8, and End of Treatment.
Description: Change in albumincorrected serum calcium from Baseline (SV2 = screening visit 2) to Week 4, Week 8, and end of treatment.
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 30
mmol/L | -0.028 (0.087)

8. Primary Outcome: Change in Albumincorrected Serum Calcium From Baseline (SV2) to Week 4, Week 8, and End of Treatment.
Description: as for outcome 7
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 26
mmol/L | 0.002 (0.087)

9. Primary Outcome: Change in Albumincorrected Serum Calcium From Baseline (SV2) to Week 4, Week 8, and End of Treatment.
Description: as for outcome 7
Time Frame: Baseline and end of treatment (up to 8 weeks)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 30
mmol/L | -0.007 (0.090)

10. Primary Outcome: Change in 24-hour Urinary Calcium Excretion From Baseline (SV2) to Week 4, Week 8, and End of Treatment.
Description: Change in 24-hour urinary calcium excretion from Baseline (SV2 = screening visit 2) to Week 4, Week 8, and end of treatment.
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: mmol/24h
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 28
mmol/24h | 0.20 (2.26)

11. Primary Outcome: Change in 24-hour Urinary Calcium Excretion From Baseline (SV2) to Week 4, Week 8, and End of Treatment.
Description: as for outcome 10
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: mmol/24h
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 22
mmol/24h | 0.06 (2.35)

12. Primary Outcome: Change in 24-hour Urinary Calcium Excretion From Baseline (SV2) to Week 4, Week 8, and End of Treatment.
Description: as for outcome 10
Time Frame: Baseline and end of treatment (up to 8 weeks)
Measure: Mean (Standard Deviation); unit: mmol/24h
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 29
mmol/24h | 0.12 (2.14)

13. Primary Outcome: Change in Urinary Calcium:Creatinine Ratio From Baseline (SV2) to Week 4, Week 8 and, End of Treatment.
Description: Change in urinary calcium:creatinine ratio from Baseline (SV2 = screening visit 2) to Week 4, Week 8 and, end of treatment.
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 28
mmol/g | -0.179 (1.848)

14. Primary Outcome: Change in Urinary Calcium:Creatinine Ratio From Baseline (SV2) to Week 4, Week 8 and, End of Treatment.
Description: as for outcome 13
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 22
mmol/g | -0.005 (2.379)

15. Primary Outcome: Change in Urinary Calcium:Creatinine Ratio From Baseline (SV2) to Week 4, Week 8 and, End of Treatment.
Description: as for outcome 13
Time Frame: Baseline and end of treatment (up to 8 weeks)
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 29
mmol/g | 0.096 (2.142)

16. Secondary Outcome: Change in Plasma PTH From Baseline (SV2) to Week 4 and Week 8
Description: Change in plasma PTH (parathyroid hormone) from Baseline (SV2 = screening visit 2) to Week 4 and Week 8
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 25
ng/L | -2.4 (15.2)

17. Secondary Outcome: Subjects With Controlled Disease (i.e., Clear or Almost Clear) According to the Investigator's Global Assessment (IGA) of Disease Severity at Weeks 2, 4, 8, and End of Treatment.
Description: Disease severity of the scalp psoriasis as assessed by the 6-point scale IGA, based on the condition of the disease at the time of evaluation. The IGA scale: 1 = clear, 2 = almost clear, 3 = mild, 4 = moderate, 5 = severe, and 6 = very severe.
Time Frame: week 2
Measure: Number; unit: percentage of participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 31
percentage of participants | 32.3

18. Secondary Outcome: Subjects With Controlled Disease (i.e., Clear or Almost Clear) According to the Investigator's Global Assessment (IGA) of Disease Severity at Weeks 2, 4, 8, and End of Treatment.
Description: Disease severity of the scalp psoriasis as assessed by the 6-point scale IGA, based on the condition of the disease at the time of evaluation.
Time Frame: week 4
Measure: Number; unit: percentage of participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 30
percentage of participants | 43.3

19. Secondary Outcome: Subjects With Controlled Disease (i.e., Clear or Almost Clear) According to the Investigator's Global Assessment (IGA) of Disease Severity at Weeks 2, 4, 8, and End of Treatment.
Description: as for outcome 18
Time Frame: week 8
Measure: Number; unit: percentage of participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 26
percentage of participants | 53.8

20. Secondary Outcome: Subjects With Controlled Disease (i.e., Clear or Almost Clear) According to the Investigator's Global Assessment (IGA) of Disease Severity at Weeks 2, 4, 8, and End of Treatment.
Description: as for outcome 18
Time Frame: End of treatment
Measure: Number; unit: percentage of participants
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 31
percentage of participants | 54.8

21. Secondary Outcome: Percentage Change in Total Sign Score (TSS; Sum of Severity Scores for Each Individual Clinical Sign, Redness, Thickness, and Scaliness) From Baseline to Weeks 2, 4, 8, and End of Treatment.
Description: Investigator assessment of scalp psoriasis lesions in terms of the three clinical signs: redness, thickness, and scaliness. Each clinical sign, a single score(ranging from 0 to 4), reflecting the average severity of all psoriatic lesions on the scalp, were determined. The sum of the three scores (redness, thickness, and scaliness) constitutes the Total Sign Score of the psoriasis on scalp, ranging from 0 (best possible outcome) to 12 points (worst possible outcome).
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 31
Percentage change | -48.0 (31.0)

22. Secondary Outcome: Percentage Change in Total Sign Score (TSS; Sum of Severity Scores for Each Individual Clinical Sign, Redness, Thickness, and Scaliness) From Baseline to Weeks 2, 4, 8, and End of Treatment.
Description: Investigator assessment of scalp psoriasis lesions in terms of the three clinical signs: redness, thickness, and scaliness. Each clinical sign, a single score (ranging from 0 to 4), reflecting the average severity of all psoriatic lesions on the scalp, were determined. The sum of the three scores (redness, thickness, and scaliness) constitutes the Total Sign Score of the psoriasis on scalp, ranging from 0 (best possible outcome) to 12 points (worst possible outcome).
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 30
percentage change | -48.8 (29.9)

23. Secondary Outcome: Percentage Change in Total Sign Score (TSS; Sum of Severity Scores for Each Individual Clinical Sign, Redness, Thickness, and Scaliness) From Baseline to Weeks 2, 4, 8, and End of Treatment.
Description: as for outcome 22
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 26
Percentage change | -57.2 (33.9)

24. Secondary Outcome: Percentage Change in Total Sign Score (TSS; Sum of Severity Scores for Each Individual Clinical Sign,Redness, Thickness, and Scaliness) From Baseline to Weeks 2, 4, 8, and End of Treatment.
Description: as for outcome 22
Time Frame: Baseline and end of treatment (up to 8 weeks)
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 31
Percentage change | -59.2 (35.4)

25. Secondary Outcome: Subjects With Controlled Disease (Defined as Clear or Very Mild) According to the Patient's Global Assessment of Disease Severity at Weeks 2, 4, 8, and End of Treatment.
Description: Disease severity of the scalp psoriasis as assessed by the 5-point scale, Patient's Global Assessment of Disease Severity, based on the condition of the disease at the time of evaluation. The scale scores are based on the following; 1 = clear, 2 = very mild, 3 = mild, 4 = moderate, 5 = severe.
Time Frame: week 2
Measure: Number; unit: % of participants w/ controlled disease
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 31
% of participants w/ controlled disease | 45.2

26. Secondary Outcome: Subjects With Controlled Disease (Defined as Clear or Very Mild) According to the Patient's Global Assessment of Disease Severity at Weeks 2, 4, 8, and End of Treatment.
Description: Disease severity of the scalp psoriasis as assessed by the 5-point scale, Patient's Global Assessment of Disease Severity, based on the condition of the disease at the time of evaluation.
Time Frame: week 4
Measure: Number; unit: % of participants w/ controlled disease
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 30
% of participants w/ controlled disease | 50.0

27. Secondary Outcome: Subjects With Controlled Disease (Defined as Clear or Very Mild) According to the Patient's Global Assessment of Disease Severity at Weeks 2, 4, 8, and End of Treatment.
Description: as for outcome 26
Time Frame: week 8
Measure: Number; unit: % of participants w/ controlled disease
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 26
% of participants w/ controlled disease | 57.7

28. Secondary Outcome: Subjects With Controlled Disease (Defined as Clear or Very Mild) According to the Patient's Global Assessment of Disease Severity at Weeks 2, 4, 8, and End of Treatment.
Description: as for outcome 26
Time Frame: End of treatment
Measure: Number; unit: % of participants w/ controlled disease
Arm/Group | LEO 80185 Gel
Number analyzed (Participants) | 31
% of participants w/ controlled disease | 58.1

ADVERSE EVENTS:
Arm/Group | LEO 80185 Gel
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 10/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 80185 Gel (N=31)
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Nasopharyngitis (Infections and infestations) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Upper respiratory tract (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators' right to publish the results of the trial, irrespective of outcome. Pubs/presentations by investigator(s) shall not be made before the results of a joint publication is public. LEO retains the right to have any publication submitted to LEO for review at least 30 days prior to this paper being submitted for publication/presentation. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.